CLINICAL TRIAL: NCT04912102
Title: High Flow Nasal Oxygen Versus Nasal Continuous Positive Airway Pressure in Obese Patients Undergoing Deep Sedation for Endoscopic Retrograde Cholangiopancreatography: A Randomized Controlled Trial
Brief Title: HFNO Versus Nasal CPAP in Obese Patients Undergoing Deep Sedation for ERCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mennat Allah Mahmoud Bakri, assisstant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HFNO Vs CPAP in ERCP
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group H (Active Comparator): Oxygen will be delvered via HFNO canula at 20 L/min, Fio2 0.4 and temperature of 37o c using Vapotherm Precision Flow.
  Interventions: Device: high flow nasal oxygen device (HFNO)
- Group M (Active Comparator): Mask group will be provided with nasal CPAP (10cmH2O) at an oxygen flow rate of 15 L/min.
  Interventions: Device: high flow nasal oxygen device (HFNO)
- Group C (Active Comparator): In the Control group, oxygen via a nasal cannula at a flow rate of 5 L/min will be delivered
  Interventions: Device: high flow nasal oxygen device (HFNO)

INTERVENTIONS:
Device: high flow nasal oxygen device (HFNO) — it is a novel technique by which heated humidified oxygen is supplied via nasal prongs at flow rates ranging from 40 to 70 L/minute. The Fio2 ranges from 0.21 to 1.0.

SUMMARY:
Endoscopic retrograde cholangio-pancreatography (ERCP) is commonly performed under deep sedation to provide amnesia, comfort, and optimal procedural conditions. However, anesthetic drugs commonly used such as midazolam and/or propofol and opioids for sedative endoscopy in clinical practice may depress normal ventilation by blunting central chemoreceptor responsiveness to CO2, and alveolar hypoventilation and predispose patients to upper airway obstruction; all of that can result in hypoxemia, hypercarbia, respiratory acidosis, hypotension, and, in rare cases, brain injury or death.(1-3)

DETAILED DESCRIPTION:
The incidence of hypoxia during ERCP with sedation has been reported to range from 16.2 to 39.2% (4) may be because ERCP procedures can be lengthy and are often performed in the prone position.(5) Hypoxemia is the most common adverse cardiopulmonary complication during sedated endoscopy and is caused by respiratory depression, airway obstruction, and decreased chest wall compliance. (2)

Obese patients are particularly at risk of upper airway obstruction and hypoxemia under sedation and may benefit from Conventional CPAP, applied nasally to improve ventilation and oxygenation during spontaneous ventilation in patients under deep sedation through maintenance of upper airway patency.(6) Recently novel techniques have been shown to be more effectively help ventilation than conventional low flow nasal oxygen. High flow nasal oxygen (HFNO) has been utilized in the intensive care setting for over 15 years. Its use in anaesthesia is rapidly increasing, providing an alternative to low flow oxygen devices during sedation for procedures such as gastroenterology, non-invasive cardiological, radiological, emergency medicine and persistent pain procedures.(1) Multiple mechanisms account for the therapeutic effects of HFNO, including a reduction in dead space, increased positive end-expiratory pressure, increased functional residual capacity, and delivery of higher inspired oxygen concentrations to the distal airways.(7) Moreover the heated and humidified HFNO provides adequate oxygenation with less drying of the upper airway mucosa, thereby improving patient comfort.(8) The use of HFNO in the gastroenterological suite had reduced critical incidents by providing high-inspired oxygen and slowing carbon dioxide rises related to respiratory depression.

Maintaining patient safety while successfully completing the procedures under sedation requires careful monitoring. Australian and New Zealand College of Anaesthetists (ANZCA) Guidelines on Monitoring during Anaesthesia, the Association of Anaesthetists of Great Britain & Ireland (AAGBI) and the American Society of Anesthesiologists Standards for Basic Anesthetic Monitoring had all emphasized the importance of monitoring exhaled Co2 during moderate to deep sedation to improve patients' safety. (9) Monitoring EtCO2 for the anesthesiologist is more superior to the pulse oximeter for immediately detecting an obstructed airway, opiate-induced apnea, or other airway problems that only much later may be detected by the pulse oximeter.(9) Unfortunately, it would be expected that the high oxygen flow rates during HFNO would severely dilute expired carbon dioxide and make sampling impossible.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective ERCP with deep sedation will be enrolled
* age 18 - 70 years old
* obesity (BMI 30-35 kg/m2)
* American Society of Anaesthesiologists' physical status classification of 1 to 3
* Anticipated duration of the procedure is > 15 minutes.

Exclusion Criteria:

* • BMI >35 kg/m2

  * Simple procedures of < 15 minutes duration.
  * untreated or unstable cardiac conditions
  * Nasal or oral disease resulting in difficulty of either nasal breathing or mouth breathing.
  * Acute or chronic respiratory disorders as asthma and chronic obstructive pulmonary disease.
  * Pregnant patients and patients having procedures with planned endotracheal intubation
  * Expected difficult intubation patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2021-10-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
A hypoxemia event | for 15 consecutive secondes
  Spo2 <92% for at least 15 consecutive seconds (we based our definition on prior studies)

SECONDARY OUTCOMES:
The lowest Spo2 reading | during the whole procedure
  the lowest spo2
Incidence of hypercapnia | before induction, 5 min after induction and then every 10 min till end of procedure
  PaCo2 will be assessed in an venous blood gas sample drawn before induction of anaesthesia and second sample 5 min. after induction and then every 10 min till the end of the procedure

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bhananker SM, Posner KL, Cheney FW, Caplan RA, Lee LA, Domino KB. Injury and liability associated with monitored anesthesia care: a closed claims analysis. Anesthesiology. 2006 Feb;104(2):228-34. doi: 10.1097/00000542-200602000-00005. PMID 16436839
- [Background] Amornyotin S. Sedation-related complications in gastrointestinal endoscopy. World J Gastrointest Endosc. 2013 Nov 16;5(11):527-33. doi: 10.4253/wjge.v5.i11.527. PMID 24255744
- [Background] Mazzeffi MA, Petrick KM, Magder L, Greenwald BD, Darwin P, Goldberg EM, Bigeleisen P, Chow JH, Anders M, Boyd CM, Kaplowitz JS, Sun K, Terrin M, Rock P. High-Flow Nasal Cannula Oxygen in Patients Having Anesthesia for Advanced Esophagogastroduodenoscopy: HIFLOW-ENDO, a Randomized Clinical Trial. Anesth Analg. 2021 Mar 1;132(3):743-751. doi: 10.1213/ANE.0000000000004837. PMID 32398433
- [Background] Wang CY, Ling LC, Cardosa MS, Wong AK, Wong NW. Hypoxia during upper gastrointestinal endoscopy with and without sedation and the effect of pre-oxygenation on oxygen saturation. Anaesthesia. 2000 Jul;55(7):654-8. doi: 10.1046/j.1365-2044.2000.01520.x. PMID 10919420
- [Background] Muller S, Prolla JC, Maguilnik I, Breyer HP. Predictive factors of oxygen desaturation of patients submitted to endoscopic retrograde cholangiopancreatography under conscious sedation. Arq Gastroenterol. 2004 Jul-Sep;41(3):162-6. doi: 10.1590/s0004-28032004000300005. Epub 2005 Jan 21. PMID 15678200
- [Background] Andrade RG, Piccin VS, Nascimento JA, Viana FM, Genta PR, Lorenzi-Filho G. Impact of the type of mask on the effectiveness of and adherence to continuous positive airway pressure treatment for obstructive sleep apnea. J Bras Pneumol. 2014 Nov-Dec;40(6):658-68. doi: 10.1590/S1806-37132014000600010. PMID 25610507
- [Background] Nishimura M. High-flow nasal cannula oxygen therapy in adults. J Intensive Care. 2015 Mar 31;3(1):15. doi: 10.1186/s40560-015-0084-5. eCollection 2015. PMID 25866645
- [Background] Greenland KB. A potential method for obtaining wave-form capnography during high flow nasal oxygen. Anaesth Intensive Care. 2019 Mar;47(2):204-206. doi: 10.1177/0310057X19836430. Epub 2019 May 1. No abstract available. PMID 31042046
- [Background] Weaver J. The latest ASA mandate: CO(2) monitoring for moderate and deep sedation. Anesth Prog. 2011 Fall;58(3):111-2. doi: 10.2344/0003-3006-58.3.111. No abstract available. PMID 21882985